CLINICAL TRIAL: NCT01857102
Title: Toric Eye Strain and Stability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5363
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2017-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- etafilcon A/etafilcon A for Astigmatism (Active Comparator): Subjects were randomized to one of two sequences of lens wear.
  Interventions: Device: etafilcon A; Device: etafilcon A for Astigmatism
- etafilcon A for Astigmatism/etafilcon A (Experimental): Subjects were randomized to one of two sequences of lens wear.
  Interventions: Device: etafilcon A; Device: etafilcon A for Astigmatism

INTERVENTIONS:
Device: etafilcon A — Soft contact lens to be worn in a daily wear, daily disposable modality for one week
Device: etafilcon A for Astigmatism — Soft contact lens to be worn by participants in a daily wear, daily disposable modality for one week.

SUMMARY:
The purpose of this study is to determine the benefits of fitting low astigmats with soft toric contact lenses versus spherical contact lenses with regard to visual comfort, eyestrain, fitting efficiency, and visual performance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have read, understand, and sign the statement of informed consent and receive a fully executed copy of the Informed Consent Form.
2. The subject must appear able and willing to adhere to the instructions set forth in this protocol.
3. The subject must be between 18 years and 45 years of age (inclusive).
4. The subject must have best-corrected Snellen visual acuity of 20/30 or better in each eye.
5. If the subject has ever worn contact lenses, the subject must be a current wearer of soft spherical contact lenses for at least 5 days/week and at least 8 hours/day during the month prior to enrollment.
6. Subjective refraction must result in a vertex-corrected astigmatic contact lens prescription requiring at least -0.75 DC but not more than -1.75 DC cylindrical contact lens correction in each eye.
7. Subjective refraction must result in a vertex-corrected spherical contact lens prescription between +0.25D to +4.00D or between-0.50D to -9.00D in each eye.
8. The subject must not have the need for presbyopic correction (i.e., they must not be using as add in spectacles or wearing multifocal or monofocal contact lenses).
9. The subject must have normal eyes with no evidence of abnormality or disease that in the opinion of the investigator would contraindicate contact lens wear.
10. The subject must have access to the internet throughout the day (either desktop and/or smartphone) and be willing to answer a web-based survey within 1 hour of receiving a text message based notification throughout the day for up to 8 days, throughout the study duration.

Exclusion Criteria:

1. Self-reported current pregnancy or lactation or plans to become pregnant during the study period (subjects who report becoming pregnant during the study will be discontinued)
2. Any previous ocular or intra-ocular surgery (e.g. radial keratotomy, PRK, LASIK, etc.)
3. Any clinically meaningful slit lamp findings contraindicating contact lens wear (e.g. greater than or equal to grade 3 finding of edema, corneal neovascularization, corneal staining, conjunctival injection, blepharitis/meibomian gland dysfunction) on the FDA classification scale or any other ocular abnormality that in the opinion of the investigator may contraindicate contact lens wear.
4. Any ocular infection
5. Current use of topical ophthalmic medications other than artificial tears/rewetting drops.
6. History of binocular vision abnormality or strabismus.
7. Any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV) by self-report.
8. Other active ocular disease that in the opinion of the investigator would contraindicate contact lens wear.
9. Employee of the investigational clinic (e.g. investigator, coordinator, technician)
10. Subject does not have a wearable pair of spectacles.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 159 (Actual)
Dates: Start 2013-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 159 subjects were enrolled in the study. Of the enrolled subjects 45 did not meet the eligibility criteria and 114 subjects were dispensed a study lens. Of the dispensed subjects 10 subjects were discontinued and 94 subjects completed the study.
Pre-assignment Details: Of those completed 24 were excluded from the analysis due to a major protocol deviation. Of the subjects that completed all study visits without a major protocol deviation, 10 subjects were classified as neophytes and 60 as habitual contact lens users.
Groups:
- Etafilcon A/ Etafilcon A for Astigmatism: Subjects that first received the etafilcon A lens and then received the etafilcon A for Astigmatism lens.
- Etafilcon A for Astigmatism/Etafilcon A: Subjects that first received the etafilcon A for Astigmatism lens and then received the etafilcon A lens.
Period: Period 1
Arm/Group | Etafilcon A/ Etafilcon A for Astigmatism | Etafilcon A for Astigmatism/Etafilcon A
Started | 58 | 56
Habitual Users | 51 | 52
Neophtyes | 7 | 4
Completed | 55 | 51
Not Completed | 3 | 5
Not completed — No longer meets Eligibility Criteria | 0 | 2
Not completed — Lost to Follow-up | 0 | 3
Not completed — Unsatisfactory Lens Fit | 1 | 0
Not completed — Unsatisfactory Visual Response | 1 | 0
Not completed — Physician Decision | 1 | 0
Period: Period 2
Arm/Group | Etafilcon A/ Etafilcon A for Astigmatism | Etafilcon A for Astigmatism/Etafilcon A
Started | 55 | 51
Habitual Users | 48 | 47
Neophytes | 7 | 4
Completed | 53 | 51
Not Completed | 2 | 0
Not completed — Lens Discomfort | 1 | 0
Not completed — Unsatisfactory Lens Fit | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population consists of all subjects that were dispensed at least one study lens.
Groups:
- Dispensed Subjects: All subjects that were dispensed at least one study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 114
Age, Continuous [Mean (Standard Deviation); unit: years]
  Habitual Users | 26.9 (4.93)
  Neophtyes | 28.5 (2.66)
  Overall | 27.1 (4.77)
Sex: Female, Male [Count of Participants; unit: Participants] — All subjects that were dispensed a study lens.
  Participants
    Female | 75
    Male | 39
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 3
  Asian | 34
  Black or African American | 18
  Native Hawaiian or Pacific Islander | 2
  White | 49
  Other | 8
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Objective Comfort Assessed by Electromyography(EMG)
Description: Electromyography (EMG) utilizes electrodes affixed to the skin below the eyelid, which measures activity of the orbital portion of the orbicularis oculi muscle. The orbital portion of the orbicularis oculi muscle pulls on the skin of the forehead, temple and cheek and draws it toward a point at the edge of the orbit. This part of the muscle is mainly under voluntary control, and it what is contracted during the process of squinting. The palpebral portion of this muscle closes the eyelids. The EMG reading was performed while the subject was wearing contact lenses in order to objectively assess eyestrain.The higher the EMG reading indicated the more the eyestrain. The original EMG data collected from a 40-second recording consisted of approximately 40,000 observations; the machine read about 1000 observations per second consecutively during 40-second recording. The original EMG reading was converted to a single data point and entered in the EDC for the analysis purpose.
Time Frame: 1 week
Population: Analysis population consists of all subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: volts
Groups:
- Etafilcon A: Subjects that received the etafilcon A lens in either the first or second period of the study.
- Etafilcon A for Astigmatism: Subjects that received the etafilcon A for Astigmatism lens in either the first or second period of the study.
Arm/Group | Etafilcon A | Etafilcon A for Astigmatism
Number analyzed (Participants) | 70 | 70
volts
  Habitual Users, N=60, N=60 | 0.082 (0.1239) | 0.047 (0.0599)
  Neophytes, N=10, N=10 | 0.085 (0.0940) | 0.257 (0.6310)

2. Primary Outcome: Visual Comfort
Description: The Visual comfort (diurnal fluctuation[DF]) scores were derived from the National Eye Institute Refractive Error Quality of Life (NEI-RQL) instruments- specifically the diurnal fluctuations sub-scale, by following the instruction given in the NEI-RQL-42 User Manual, Version 1.0. The NEI-RQL is a validated patient reported outcome questionnaire to assess the impact of refractive correction on vision specifically to quality of life. This survey consisted of 42 items used to develop 13 subscales: clarity of vision, expectations, near vision, far vision, diurnal fluctuations, activity limitations, glare, symptoms, dependence on correction, worry, suboptimal correction, appearance, and satisfaction with correction. An overall score is calculated by averaging the subscales. The overall scores can take on values of 0 to 100. Higher scores indicate better outcomes
Time Frame: 1-week follow-up
Population: The analysis population consists of all subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Etafilcon A: Subjects that received the etafilcon A lens during the first or second period of the study.
- Etafilcon A for Astigmatism: Subjects that received etafilcon A for Astigmatism lens in either the first or second period of the study.
Arm/Group | Etafilcon A | Etafilcon A for Astigmatism
Number analyzed (Participants) | 70 | 70
units on a scale
  Habitual Users, N=60, N=60 | 72.8 (24.94) | 80.6 (19.41)
  Nepohytes, N=10, N=10 | 70.4 (21.29) | 72.5 (23.02)

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 1 month per subject.
Arm/Group | Etafilcon A | Etafilcon A for Astigmatism
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/114
Other Adverse Events (participants affected / at risk) | 0/114 | 0/114

LIMITATIONS AND CAVEATS:
Data collected on Neophyte population was for exploratory purpose only. The study was not powered to show differences in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days